CLINICAL TRIAL: NCT06183710
Title: Adjunctive Contingency Management to Incentivise Adherence to Treatment in Alcohol-related Liver Disease: a Mixed-methods Study
Brief Title: Contingency Management to Incentivise Treatment Adherence in Alcohol-related Liver Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRAS ID 314351
Record Dates: First submitted 2023-12-04; First posted 2023-12-27 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Alcohol-related Liver Disease
Keywords: Contingency management; Alcohol-use Disorder; Psychosocial intervention; Treatment adherence
MeSH Terms: conditions — Alcoholism; Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: Prospective, individually randomized pilot trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated care only (control group) (No Intervention): The integrated care comprises of standard treatment offered at the Integrated Treatment Clinic at King's College Hospital and includes addiction and liver follow-up as well as facilitation of psychosocial sessions
- Integrated care + CM (Experimental): The integrated care comprises of standard treatment offered at the Integrated Treatment Clinic at King's College Hospital and includes addiction and liver follow-up as well as facilitation of psychosocial sessions. The adjunctive CM aims to reinforce attendance to integrated alcohol and liver care services from KCH over the course of 3 months
  Interventions: Behavioral: Contingency management

INTERVENTIONS:
Behavioral: Contingency management — Psychosocial intervention
  Arms: Integrated care + CM

SUMMARY:
A sample of 30 alcohol-related liver disease patients will be recruited through consecutive sampling, facilitated through the Alcohol Care Team, which will identify potential participants to the study that have been referred to the team.

Patients will be randomised either to the control or intervention group. In the control group, patients will receive outpatient integrated liver care (hepatology, psychosocial and addiction follow-ups). In the intervention group, a contingency management intervention will be delivered in addition to integrated care.

DETAILED DESCRIPTION:
A sample of 30 ARLD patients will be recruited through consecutive sampling, facilitated through the ACT, who will identify potential participants to the study that have been referred to the team. The ACT will give service users a study advert and patient information sheet (PIS). If consented, the contact details will be passed on to the research team, who will contact potential participants. A maximum of three attempts to contact a participant will be made at each planned follow-up point (3 and 6 months).

Following referral to the study, the research student will contact the potential participant via telephone to discuss the study. The purpose of the call is to provide further details of the research, confirm whether the service user wishes to take part in the research and provide a Patient Information Sheet (PIS). The research student will allow the potential participant to clarify any initial questions related to the research and proceed to arrange an initial assessment appointment. This appointment will be set at least 24 hours after the service user receives the PIS to allow for further consideration.

When a potential participant is identified and referred to the ACT while in the emergency department, the ACT clinician will discuss the study with the patient and provide the PIS. The point at which the study is discussed with the patient may vary. This will be assessed on an individual basis by the ACT clinician, to prevent approaching patients prematurely, or if they are in distress/clinically unstable. Patients will not be approached by clinical staff about taking part in the study if they are in distress or clinically unstable.

If the patient agrees, the contact details will be passed to the research team, who will follow up to confirm interest in the study and obtain informed consent. This contact attempt is to be made at least 24 hours after the potential participant receives the study PIS.

Following study enrolment, subjects will be randomised to either:

Treatment arm 1: Integrated care only (control group) OR Treatment arm 2: Integrated care + CM (intervention group). The integrated care comprises standard treatment offered at the Integrated Treatment Clinic at King's College Hospital and includes addiction and liver follow-up as well as facilitation of psychosocial sessions. The adjunctive CM aims to reinforce attendance to integrated alcohol and liver care services from KCH for 3 months, with follow-up times at 3- and 6-months.

The use of vouchers, redeemable for goods other than alcohol or tobacco, to reward a specific behaviour is effective and regarded as being easier to implement in the NHS. The participant's attendance will be monitored by liaising with the involved treatment services (administrative task), and the incentive will be delivered by the research team, hence not interfering with the clinician's daily workflow. After confirming the attendance, the participant will be notified via text message of the awarded voucher, the number of sessions attended and the total prize value to date, and the total prize amount to be awarded by the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old or above.
2. Able to communicate in English independently.
3. Formal diagnosis of ARLD in line with ICD-10 K70 codes (fatty liver, hepatitis, fibrosis, sclerosis, cirrhosis, hepatic failure, unspecified liver disease) upon discharge following acute liver disease episode.
4. Formal diagnosis of AD in line with ICD-10 F10.2 codes.
5. Attending South London liver services (King's Health Partners).
6. Able and willing to provide informed consent.
7. Able and willing to participate in study.
8. Owning a mobile phone.

Exclusion Criteria:

1. Less than 18 years old.
2. Current dependence on other substances other than alcohol, tobacco, or cannabis.
3. Inability to communicate in English independently.
4. Being pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility rates | 1 year
  Quantitative data: eligibility and consent rates (number and percentage of screened patients who are eligible for inclusion in the study, number and percentage of eligible patients who consent to participate), recruitment rate (number of patients recruited each week over the recruitment period), intervention compliance (number and percentage of intervention sessions delivered to each of the enrolled participants) follow-up rates (number and percentage of participants followed up for research interview at 3 and 6-month follow-ups), drop-out rate (number and percentage of participants dropping out if assigned to control group)
Acceptability | 1 year
  Qualitative data (in-depth interviews): acceptability of CM intervention, perceived experience, treatment experience Quantitative data: Theoretical Framework for Acceptability survey (descriptive statistics)

CONTACTS AND LOCATIONS:
Overall Officials: Colin Drummond, Principal Investigator — King's College London
Locations (1):
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No